CLINICAL TRIAL: NCT03672175
Title: A Phase 3, Multicenter, Double-Blind, Randomized, Placebo-Controlled Study Evaluating the Efficacy of SAGE-217 in the Treatment of Adult Subjects With Major Depressive Disorder
Brief Title: A Study to Evaluate the Efficacy of SAGE-217 in the Treatment of Adult Participants With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 217-MDD-301
Record Dates: First submitted 2018-09-12; First posted 2018-09-14 (Actual); Results first posted 2022-11-10 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — zuranolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SAGE-217 Matched Placebo (Placebo Comparator): Participants self-administered SAGE-217 matched placebo capsules, orally, once daily in the evening with food for 14 days.
  Interventions: Drug: Placebo
- SAGE-217 20 mg (Experimental): Participants self-administered SAGE-217 20 milligrams (mg) capsules, orally, once daily in the evening with food for 14 days.
  Interventions: Drug: SAGE-217
- SAGE-217 30 mg (Experimental): Participants self-administered SAGE-217 30 mg capsules, orally, once daily in the evening with food for 14 days.
  Interventions: Drug: SAGE-217

INTERVENTIONS:
Drug: SAGE-217 — SAGE-217 hard gelatin capsules.
  Arms: SAGE-217 20 mg; SAGE-217 30 mg
Drug: Placebo — SAGE-217 matched placebo hard gelatin capsules.
  Arms: SAGE-217 Matched Placebo

SUMMARY:
This study is a phase 3, multicenter, double-blind, randomized, placebo-controlled study evaluating the efficacy of SAGE-217 in the treatment of adult participants with major depressive disorder (MDD).

DETAILED DESCRIPTION:
This study was previously posted by Sage Therapeutics. In November 2023, sponsorship of the trial was transferred to Biogen.

ELIGIBILITY:
Inclusion Criteria:

1. Participant had a diagnosis of MDD with symptoms that had been present for at least a 4-week period.
2. Participant had a Montgomery-Åsberg Depression Rating Scale (MADRS) total score of ≥32 and a 17-item Hamilton Rating Scale for Depression (HAM-D) total score ≥22 at screening and Day 1 (prior to dosing).

Exclusion Criteria:

1. Participant had active psychosis.
2. Participant had attempted suicide associated with the current episode of MDD.
3. Participant had a medical history of bipolar disorder, schizophrenia, and/or schizoaffective disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 581 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2019-09-24 (Actual); Study Completion 2020-03-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (47):
- United States (47):
  - Sage Investigational Site, Rogers, Arkansas
  - Sage Investigational Site, Bellflower, California
  - Sage Investigational Site, Garden Grove, California
  - Sage Investigational Site, Glendale, California
  - Sage Investigational Site, National City, California
  - Sage Investigational Site, Oakland, California
  - Sage Investigational Site, Oceanside, California
  - Sage Investigational Site, Orange, California
  - Sage Investigational Site, Pico Rivera, California
  - Sage Investigational Site, Redlands, California
  - Sage Investigational Site, San Diego, California
  - Sage Investigational Site, Sherman Oaks, California
  - Sage Investigational Site, Temecula, California
  - Sage Investigational Site, Coral Springs, Florida
  - Sage Investigational Site, Hollywood, Florida
  - Sage Investigational Site, Jacksonville, Florida
  - Sage Investigational Site, Lauderhill, Florida
  - Sage Investigational Site, Maitland, Florida
  - Sage Investigational Site, North Miami, Florida
  - Sage Investigational Site, Orange City, Florida
  - Sage Investigational Site, Orlando, Florida
  - Sage Investigational Site, Atlanta, Georgia
  - Site Investigational Site, Decatur, Georgia
  - Sage Investigational Site, Skokie, Illinois
  - Sage Investigational Site, Pikesville, Maryland
  - Sage Investigational Site, Flowood, Mississippi
  - Sage Investigational Site, O'Fallon, Missouri
  - Sage Investigational Site, St Louis, Missouri
  - Sage Investigational Site, Las Vegas, Nevada
  - Sage Investigational Site, Berlin, New Jersey
  - Sage Investigational Site, Jamaica, New York
  - Sage Investigational Site, Rochester, New York
  - Sage Investigational Site, Charlotte, North Carolina
  - Sage Investigational Site, Cincinnati, Ohio
  - Sage Investigational Site, Dayton, Ohio
  - Sage Investigational Site, North Canton, Ohio
  - Sage Investigational Site, Oklahoma City, Oklahoma
  - Sage Investigational Site, Portland, Oregon
  - Sage Investigational Site, Allentown, Pennsylvania
  - Sage Investigational Site, Charleston, South Carolina
  - Sage Investigational Site, Memphis, Tennessee
  - Sage Investigational Site, Austin, Texas
  - Sage Investigational Site, Bellaire, Texas
  - Sage Investigational Site, DeSoto, Texas
  - Sage Investigational Site, Richardson, Texas
  - Sage Investigational Site, Wichita Falls, Texas
  - Sage Investigational Site, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

REFERENCES:
- [Derived] Clayton AH, Lasser R, Nandy I, Sankoh AJ, Jonas J, Kanes SJ. Zuranolone in Major Depressive Disorder: Results From MOUNTAIN-A Phase 3, Multicenter, Double-Blind, Randomized, Placebo-Controlled Trial. J Clin Psychiatry. 2023 Feb 20;84(2):22m14445. doi: 10.4088/JCP.22m14445. PMID 36811520
- See also: Related Info — http://www.sagerx.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in the study at 55 centers in the United States from 19 November 2018 to 17 March 2020.
Pre-assignment Details: A total of 1327 participants were screened of which 581 were randomized and 570 were dosed. This study consisted of up to a 28-day screening period, a 14-day treatment period, a 28-day follow-up (FU) period, and an extended FU period through Day 182 (6 months following the last dose).
Groups:
- SAGE-217 20 mg: Participants self-administered SAGE-217 20 mg capsules, orally, once daily in the evening with food for 14 days.
Period: Treatment Period (Days 1 to 14)
Arm/Group | SAGE-217 Matched Placebo | SAGE-217 20 mg | SAGE-217 30 mg
Started | 193 | 194 | 194
Safety Set (Safety Set included all participants who were administered investigational product (IP) [SAGE-217 20 mg, SAGE-217 30 mg, or SAGE-217 matched placebo].) | 190 | 188 | 192
Modified Full Analysis Set (mFAS) (mFAS included all randomized participants with valid baseline Hamilton Rating Scale for Depression (HAM-D) and at least 1 post-baseline HAM-D evaluation, with a total HAM-D score of at least 22 at baseline.) | 157 | 159 | 166
Completed | 182 | 180 | 185
Not Completed | 11 | 14 | 9
Not completed — Withdrawal by Subject | 6 | 6 | 4
Not completed — Lost to Follow-up | 2 | 2 | 3
Not completed — Randomized but not Treated | 3 | 6 | 2
Period: FU Period (Days 15 to 42)
Arm/Group | SAGE-217 Matched Placebo | SAGE-217 20 mg | SAGE-217 30 mg
Started | 182 | 180 | 185
Completed | 178 | 170 | 178
Not Completed | 4 | 10 | 7
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Lost to Follow-up | 3 | 6 | 2
Not completed — Withdrawal by Subject | 1 | 4 | 4
Period: Extended FU Period (Days 43 to 182)
Arm/Group | SAGE-217 Matched Placebo | SAGE-217 20 mg | SAGE-217 30 mg
Started | 178 | 170 | 178
Extended FU Safety Set (Extended FU Safety Set included all participants in the Safety Set of treatment period who consented or reconsented to participate in the study in the 6-month FU period.) | 129 | 127 | 131
Completed | 141 | 131 | 141
Not Completed | 37 | 39 | 37
Not completed — Adverse Event | 5 | 3 | 3
Not completed — Lost to Follow-up | 6 | 8 | 7
Not completed — Non-compliance with Study Drug | 1 | 0 | 1
Not completed — Reason not Specified | 3 | 4 | 3
Not completed — Physician Decision | 4 | 0 | 2
Not completed — Withdrawal by Subject | 18 | 24 | 21

BASELINE CHARACTERISTICS:
Population: Safety Set included all participants who were administered IP.
Groups:
- Total: Total of all reporting groups
Arm/Group | SAGE-217 Matched Placebo | SAGE-217 20 mg | SAGE-217 30 mg | Total
Number analyzed (Participants) | 190 | 188 | 192 | 570
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (12.25) | 42.5 (12.10) | 42.5 (11.82) | 42.1 (12.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130 | 131 | 137 | 398
  Male | 60 | 57 | 55 | 172
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30 | 35 | 29 | 94
  Not Hispanic or Latino | 160 | 153 | 163 | 476
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 118 | 119 | 108 | 345
  Race: Black or African-American | 60 | 64 | 75 | 199
  Race: Asian | 5 | 4 | 3 | 12
  Race: More than One Race | 5 | 1 | 4 | 10
  Race: Other | 1 | 0 | 2 | 3
  Race: American-Indian or Alaska Native | 1 | 0 | 0 | 1
17-item HAM-D Total Score [Mean (Full Range); unit: score on a scale] — The HAM-D total score comprises a sum of the 17 individual item scores. 8 items scored in a range of 0 to 2 include: Insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. The following 9 items are scored in a range of 0 to 4: Agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety (psychic and somatic), and hypochondriasis. Total HAM-D score can range from 0 to 52, and higher scores indicate severe depression. Population: mFAS included all randomized participants with valid baseline HAM-D and at least 1 post-baseline HAM-D evaluation, with a total HAM-D score of at least 22 at baseline.
  score on a scale
    number analyzed (Participants) | 157 | 159 | 166 | 482
    (all) | 25.8 [22 to 36] | 25.8 [22 to 33] | 25.9 [22 to 35] | 25.8 [22 to 36]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the 17-item HAM-D Total Score at Day 15
Description: The 17-item HAM-D is used to rate the severity of depression in participants who were already diagnosed as depressed. The HAM-D total score comprises a sum of the 17 individual item scores. 8 items scored in a range of 0 to 2 include: Insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. The following 9 items are scored in a range of 0 to 4: Agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety (psychic and somatic), and hypochondriasis. Total HAM-D score can range from 0 to 52, and higher scores indicate severe depression. A negative change from baseline indicates less depression.
Time Frame: Baseline (BL), Day 15
Population: mFAS included all randomized participants with valid baseline HAM-D and at least 1 post-baseline HAM-D evaluation, with a total HAM-D score of at least 22 at baseline. Here, "Overall number of participants analyzed" is the number of participants with data available for analyses.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | SAGE-217 Matched Placebo | SAGE-217 20 mg | SAGE-217 30 mg
Number analyzed (Participants) | 141 | 152 | 153
score on a scale | -11.1 (0.59) | -11.5 (0.62) | -12.5 (0.68)
Statistical Analysis 1: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Mixed effect model for repeated measures (MMRM); Test type: Superiority; p = 0.6638, MMRM — MMRM was used for analysis with change from BL in HAM-D total score as dependent variable; treatment, BL HAM-D total score, antidepressant use, assessment time point, time point-by-treatment interaction as explanatory variables and fixed effects; Least Square (LS) Mean Difference = -0.4, 95% CI 2-sided [-2.0 to 1.3], Standard Error of Mean 0.85
Statistical Analysis 2: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Test type: Superiority; p = 0.1158, MMRM — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -1.4, 95% CI 2-sided [-3.1 to 0.3], Standard Error of Mean 0.89

2. Secondary Outcome: Change From Baseline in Clinical Global Impression - Severity (CGI-S) Score at Day 15
Description: The CGI-S uses a 7-point Likert scale to rate the severity of the participant's illness relative to the clinician's past experience with participants who had the same diagnosis. Considering total clinical experience, a participant was assessed on severity of mental illness at the time of rating as 1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; and 7=extremely ill. A higher score indicates extreme illness/more severity. A negative change from baseline indicates less severe illness.
Time Frame: Baseline, Day 15
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | SAGE-217 Matched Placebo | SAGE-217 20 mg | SAGE-217 30 mg
Number analyzed (Participants) | 141 | 151 | 152
score on a scale | -1.5 (0.10) | -1.6 (0.11) | -1.7 (0.11)
Statistical Analysis 1: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Test type: Superiority; p = 0.6905, MMRM — MMRM was used for the analysis. Treatment, BL CGI-S score, BL antidepressant use, assessment time point, and time point-by-treatment interaction were included in the model and were treated as fixed effects; LS Mean Difference = -0.1, 95% CI 2-sided [-0.4 to 0.2], Standard Error of Mean 0.15
Statistical Analysis 2: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Test type: Superiority; p = 0.1082, MMRM — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.2, 95% CI 2-sided [-0.5 to 0.1], Standard Error of Mean 0.15

3. Secondary Outcome: Change From Baseline in the 17-item HAM-D Total Score
Description: as for outcome 1
Time Frame: Baseline, Days 3, 8, 42, and 182
Population: mFAS included all randomized participants with valid baseline HAM-D and at least 1 post-baseline HAM-D evaluation, with a total HAM-D score of at least 22 at baseline. Here, "Overall number of participants analyzed" is the number of participants with data available for analyses. "Number analyzed" is the number of participants evaluable for this outcome measure at specified time points.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | SAGE-217 Matched Placebo | SAGE-217 20 mg | SAGE-217 30 mg
Number analyzed (Participants) | 157 | 158 | 163
score on a scale
  Change from Baseline at Day 3 | -6.7 (0.46) | -7.1 (0.48) | -8.3 (0.47)
  Change from Baseline at Day 8: number analyzed (Participants) | 152 | 155 | 160
  Change from Baseline at Day 8 | -7.8 (0.53) | -8.4 (0.54) | -9.9 (0.60)
  Change from Baseline at Day 42: number analyzed (Participants) | 135 | 140 | 136
  Change from Baseline at Day 42 | -11.7 (0.64) | -11.5 (0.70) | -11.9 (0.67)
  Change from Baseline at Day 182: number analyzed (Participants) | 88 | 77 | 87
  Change from Baseline at Day 182 | -13.2 (0.74) | -13.4 (0.83) | -13.9 (0.72)
Statistical Analysis 1: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 3; Test type: Superiority; p = 0.5725, MMRM — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -0.4, 95% CI 2-sided [-1.7 to 0.9], Standard Error of Mean 0.65
Statistical Analysis 2: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 3; Test type: Superiority; p = 0.0160, MMRM — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -1.5, 95% CI 2-sided [-2.8 to -0.3], Standard Error of Mean 0.64
Statistical Analysis 3: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 8; Test type: Superiority; p = 0.4450, MMRM — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -0.6, 95% CI 2-sided [-2.1 to 0.9], Standard Error of Mean 0.75
Statistical Analysis 4: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 8; Test type: Superiority; p = 0.0081, MMRM — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -2.1, 95% CI 2-sided [-3.6 to -0.5], Standard Error of Mean 0.79
Statistical Analysis 5: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 42; Test type: Superiority; p = 0.8219, MMRM — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = 0.2, 95% CI 2-sided [-1.6 to 2.1], Standard Error of Mean 0.95
Statistical Analysis 6: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 42; Test type: Superiority; p = 0.8166, MMRM — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -0.2, 95% CI 2-sided [-2.0 to 1.6], Standard Error of Mean 0.92
Statistical Analysis 7: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 182; Test type: Superiority; p = 0.9000, MMRM — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-2.3 to 2.0], Standard Error of Mean 1.11
Statistical Analysis 8: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 182; Test type: Superiority; p = 0.5004, MMRM — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -0.7, 95% CI 2-sided [-2.7 to 1.3], Standard Error of Mean 1.03

4. Secondary Outcome: Number of Participants Achieving HAM-D Response
Description: HAM-D response is defined as a ≥50% reduction in HAM-D score from baseline. The HAM-D total score comprises a sum of the 17 individual item scores. 8 items scored in a range of 0 to 2 include: Insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. The following 9 items are scored in a range of 0 to 4: Agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety (psychic and somatic), and hypochondriasis. Total HAM-D score can range from 0 to 52, and higher scores indicate severe depression.
Time Frame: Days 15, 42, and 182
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | SAGE-217 Matched Placebo | SAGE-217 20 mg | SAGE-217 30 mg
Number analyzed (Participants) | 141 | 152 | 153
Participants
  Day 15 | 60 | 65 | 77
  Day 42: number analyzed (Participants) | 135 | 140 | 136
  Day 42 | 56 | 59 | 59
  Day 182: number analyzed (Participants) | 88 | 77 | 87
  Day 182 | 51 | 39 | 51
Statistical Analysis 1: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 15: Generalized estimating equation (GEE); Test type: Superiority; p = 0.8903, GEE — GEE for binary response model, with factors for treatment, BL HAM-D total score, stratification factor (anti-depressant use at BL), assessment time point, and time point-by-treatment interaction were used for analysis; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.65 to 1.63]
Statistical Analysis 2: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 15; Test type: Superiority; p = 0.1207, GEE — [p-value comment as in outcome 4, analysis 1]; Odds Ratio (OR) = 1.43, 95% CI 2-sided [0.91 to 2.25]
Statistical Analysis 3: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 42; Test type: Superiority; p = 0.7897, GEE — [p-value comment as in outcome 4, analysis 1]; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.67 to 1.70]
Statistical Analysis 4: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 42; Test type: Superiority; p = 0.6837, GEE — [p-value comment as in outcome 4, analysis 1]; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.69 to 1.76]
Statistical Analysis 5: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 182; Test type: Superiority; p = 0.6602, GEE — [p-value comment as in outcome 4, analysis 1]; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.51 to 1.53]
Statistical Analysis 6: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 182; Test type: Superiority; p = 0.9268, GEE — [p-value comment as in outcome 4, analysis 1]; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.56 to 1.69]

5. Secondary Outcome: Number of Participants Achieving HAM-D Remission
Description: HAM-D remission is defined as HAM-D total score ≤7. The HAM-D total score comprises a sum of the 17 individual item scores. 8 items scored in a range of 0 to 2 include: Insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. The following 9 items are scored in a range of 0 to 4: Agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety (psychic and somatic), and hypochondriasis. Total HAM-D score can range from 0 to 52, and higher scores indicate severe depression.
Time Frame: Days 15, 42, and 182
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | SAGE-217 Matched Placebo | SAGE-217 20 mg | SAGE-217 30 mg
Number analyzed (Participants) | 141 | 152 | 153
Participants
  Day 15 | 33 | 35 | 48
  Day 42: number analyzed (Participants) | 135 | 140 | 136
  Day 42 | 35 | 39 | 33
  Day 182: number analyzed (Participants) | 88 | 77 | 87
  Day 182 | 32 | 29 | 34
Statistical Analysis 1: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 15; Test type: Superiority; p = 0.8245, GEE — [p-value comment as in outcome 4, analysis 1]; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.62 to 1.83]
Statistical Analysis 2: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 15; Test type: Superiority; p = 0.0756, GEE — [p-value comment as in outcome 4, analysis 1]; Odds Ratio (OR) = 1.59, 95% CI 2-sided [0.95 to 2.67]
Statistical Analysis 3: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 42; Test type: Superiority; p = 0.5309, GEE — [p-value comment as in outcome 4, analysis 1]; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.70 to 2.01]
Statistical Analysis 4: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 42; Test type: Superiority; p = 0.9085, GEE — [p-value comment as in outcome 4, analysis 1]; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.56 to 1.66]
Statistical Analysis 5: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 182; Test type: Superiority; p = 0.3476, GEE — [p-value comment as in outcome 4, analysis 1]; Odds Ratio (OR) = 1.34, 95% CI 2-sided [0.73 to 2.44]
Statistical Analysis 6: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 182; Test type: Superiority; p = 0.2060, GEE — [p-value comment as in outcome 4, analysis 1]; Odds Ratio (OR) = 1.45, 95% CI 2-sided [0.82 to 2.57]

6. Secondary Outcome: Number of Participants Achieving Clinical Global Impression - Improvement (CGI-I) Response at Day 15
Description: CGI-I response is defined as a CGI-I score of very much improved or much improved. The CGI-I employs a 7-point Likert scale to measure the overall improvement in the participant's condition post-treatment. The Investigator rated the participant's total improvement whether or not it was due entirely to drug treatment. Response choices included: 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, and 7=very much worse.
Time Frame: Day 15
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SAGE-217 Matched Placebo | SAGE-217 20 mg | SAGE-217 30 mg
Number analyzed (Participants) | 141 | 151 | 152
Participants | 65 | 71 | 84
Statistical Analysis 1: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Test type: Superiority; p = 0.8303, GEE — GEE for binary response model, with factors for treatment, CGI-S BL score, anti-depressant use at BL, assessment time point, and time point-by-treatment interaction were used for analysis; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.67 to 1.65]
Statistical Analysis 2: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Test type: Superiority; p = 0.1199, GEE — [p-value comment as in outcome 6, analysis 1]; Odds Ratio (OR) = 1.43, 95% CI 2-sided [0.91 to 2.24]

7. Secondary Outcome: Change From Baseline in Hamilton Anxiety Rating Scale (HAM-A) Total Score at Day 15
Description: The 14-item HAM-A is used to rate the severity of symptoms of anxiety. Each of the 14 items is defined by a series of symptoms and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). Scoring for HAM-A is calculated by assigning scores of 0 (not present) to 4 (very severe) to each item. Total HAM-A score is calculated as the sum of the 14 individual item scores with a total score range of 0 to 56, where the score of <17 indicates mild severity, 18 to 24 indicates mild to moderate severity, and 25 to 30 indicates moderate to severe severity. A negative change from baseline indicates less severe symptoms.
Time Frame: Baseline, Day 15
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | SAGE-217 Matched Placebo | SAGE-217 20 mg | SAGE-217 30 mg
Number analyzed (Participants) | 141 | 151 | 153
score on a scale | -8.7 (0.49) | -9.1 (0.54) | -9.4 (0.53)
Statistical Analysis 1: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Test type: Superiority; p = 0.5021, MMRM — MMRM with treatment, BL HAM-A total score, anti-depressant use at BL (Yes or No), assessment time point, and time point-by-treatment interaction as fixed effects were used for analysis; LS Mean Difference = -0.5, 95% CI 2-sided [-1.9 to 0.9], Standard Error of Mean 0.71
Statistical Analysis 2: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Test type: Superiority; p = 0.2868, MMRM — [p-value comment as in outcome 7, analysis 1]; LS Mean Difference = -0.7, 95% CI 2-sided [-2.1 to 0.6], Standard Error of Mean 0.70

8. Secondary Outcome: Change From Baseline in the Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score at Day 15
Description: The MADRS is a 10-item diagnostic questionnaire used to measure the severity of depressive episodes in participants with mood disorders. Each item is rated on a 7-point scale from 0 (no symptoms) to 6 (symptoms of maximum severity). Total MADRS score, calculated as the sum of the 10 individual items, ranges from 0 to 60 with a higher score indicating more depression. A negative change from baseline indicates less severe symptoms.
Time Frame: Baseline, Day 15
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | SAGE-217 Matched Placebo | SAGE-217 20 mg | SAGE-217 30 mg
Number analyzed (Participants) | 141 | 152 | 153
score on a scale | -16.0 (0.93) | -16.7 (1.00) | -18.0 (1.03)
Statistical Analysis 1: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Test type: Superiority; p = 0.5987, MMRM — MMRM with treatment, BL MADRS total score, anti-depressant use at BL, assessment time point, and time point-by-treatment interaction as fixed effects were used for analysis; LS Mean Difference = -0.7, 95% CI 2-sided [-3.4 to 1.9], Standard Error of Mean 1.35
Statistical Analysis 2: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Test type: Superiority; p = 0.1443, MMRM — [p-value comment as in outcome 8, analysis 1]; LS Mean Difference = -2.0, 95% CI 2-sided [-4.7 to 0.7], Standard Error of Mean 1.36

9. Secondary Outcome: Change From Baseline in HAM-D Core Subscale Score
Description: The 17-item HAM-D is used to rate the severity of depression in participants who were already diagnosed as depressed. HAM-D subscale scores are calculated as the sum of the items comprising each subscale. The core subscale score is the sum of the following symptom scores, scored in a range of 0 to 4: Depressed mood, feelings of guilt, suicide, work and activities, and retardation. Total HAM-D core subscale scores were transformed to a scale of 0 to 100. Higher scores indicate more severe depression. A negative change from baseline indicates less depression.
Time Frame: Baseline, Days 15, and 42
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | SAGE-217 Matched Placebo | SAGE-217 20 mg | SAGE-217 30 mg
Number analyzed (Participants) | 141 | 152 | 153
score on a scale
  Change from Baseline at Day 15 | -21.7 (1.33) | -21.3 (1.31) | -22.6 (1.38)
  Change from Baseline at Day 42: number analyzed (Participants) | 135 | 140 | 136
  Change from Baseline at Day 42 | -23.1 (1.36) | -22.4 (1.44) | -23.6 (1.40)
Statistical Analysis 1: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 15; Test type: Superiority; p = 0.8499, MMRM — MMRM with treatment, BL HAM-D core subscale score, anti-depressant use at BL, assessment time point, and time point-by-treatment interaction as fixed effects were used for analysis; LS Mean Difference = 0.4, 95% CI 2-sided [-3.3 to 4.0], Standard Error of Mean 1.87
Statistical Analysis 2: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 15; Test type: Superiority; p = 0.6265, MMRM — [p-value comment as in outcome 9, analysis 1]; LS Mean Difference = -0.9, 95% CI 2-sided [-4.6 to 2.8], Standard Error of Mean 1.88
Statistical Analysis 3: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 42; Test type: Superiority; p = 0.7418, MMRM — [p-value comment as in outcome 9, analysis 1]; LS Mean Difference = 0.7, 95% CI 2-sided [-3.2 to 4.5], Standard Error of Mean 1.97
Statistical Analysis 4: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 42; Test type: Superiority; p = 0.7837, MMRM — [p-value comment as in outcome 9, analysis 1]; LS Mean Difference = -0.5, 95% CI 2-sided [-4.3 to 3.3], Standard Error of Mean 1.94

10. Secondary Outcome: Change From Baseline in HAM-D Anxiety Subscale Score
Description: The 17-item HAM-D is used to rate the severity of depression in participants who were already diagnosed as depressed. HAM-D subscale scores are calculated as the sum of the items comprising each subscale. The anxiety subscale score is the sum of the following symptom scores: Anxiety (psychic and somatic) [scored in a range of 0 to 4], somatic symptoms (gastrointestinal and general) [scored in a range of 0 to 2], hypochondriasis [scored in a range of 0 to 4], and loss of weight [scored in a range of 0 to 2]. Total HAM-D anxiety subscale scores were transformed to a scale of 0 to 100. Higher scores indicate more severe depression/anxiety. A negative change from baseline indicates less depression.
Time Frame: Baseline, Days 15, and 42
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | SAGE-217 Matched Placebo | SAGE-217 20 mg | SAGE-217 30 mg
Number analyzed (Participants) | 141 | 152 | 153
score on a scale
  Change from Baseline at Day 15 | -19.4 (1.19) | -20.1 (1.28) | -22.1 (1.30)
  Change from Baseline at Day 42: number analyzed (Participants) | 135 | 140 | 136
  Change from Baseline at Day 42 | -22.0 (1.27) | -20.7 (1.38) | -21.7 (1.29)
Statistical Analysis 1: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 15; Test type: Superiority; p = 0.6848, MMRM — MMRM with treatment, BL HAM-D anxiety subscale score, anti-depressant use at BL, assessment time point, and time point-by-treatment interaction as fixed effects were used for analysis; LS Mean Difference = -0.7, 95% CI 2-sided [-4.1 to 2.7], Standard Error of Mean 1.74
Statistical Analysis 2: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 15; Test type: Superiority; p = 0.1100, MMRM — [p-value comment as in outcome 10, analysis 1]; LS Mean Difference = -2.7, 95% CI 2-sided [-6.1 to 0.6], Standard Error of Mean 1.72
Statistical Analysis 3: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 42; Test type: Superiority; p = 0.5090, MMRM — [p-value comment as in outcome 10, analysis 1]; LS Mean Difference = 1.2, 95% CI 2-sided [-2.4 to 4.9], Standard Error of Mean 1.86
Statistical Analysis 4: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 42; Test type: Superiority; p = 0.8948, MMRM — [p-value comment as in outcome 10, analysis 1]; LS Mean Difference = 0.2, 95% CI 2-sided [-3.2 to 3.7], Standard Error of Mean 1.77

11. Secondary Outcome: Change From Baseline in HAM-D Bech-6 Subscale Score
Description: The 17-item HAM-D is used to rate the severity of depression in participants who were already diagnosed as depressed. HAM-D subscale scores are calculated as the sum of the items comprising each subscale. The Bech-6 subscale score is the sum of the following symptom scores, scored in a range of 0 to 4: Depressed mood, feelings of guilt, work and activities, retardation, anxiety psychic, and somatic symptoms general. Total HAM-D Bech-6 subscale scores were transformed to a scale of 0 to 100. Higher scores indicate more severe depression. A negative change from baseline indicates less depression.
Time Frame: Baseline, Days 15, and 42
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | SAGE-217 Matched Placebo | SAGE-217 20 mg | SAGE-217 30 mg
Number analyzed (Participants) | 141 | 152 | 153
score on a scale
  Change from Baseline at Day 15 | -26.2 (1.57) | -26.3 (1.62) | -28.7 (1.70)
  Change from Baseline at Day 42: number analyzed (Participants) | 135 | 140 | 136
  Change from Baseline at Day 42 | -28.0 (1.66) | -27.4 (1.77) | -28.7 (1.70)
Statistical Analysis 1: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 15; Test type: Superiority; p = 0.9591, MMRM — MMRM with treatment, BL HAM-D Bech-6 subscale score, anti-depressant use at BL, assessment time point, and time point-by-treatment interaction as fixed effects were used for analysis; LS Mean Difference = -0.1, 95% CI 2-sided [-4.5 to 4.3], Standard Error of Mean 2.25
Statistical Analysis 2: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 15; Test type: Superiority; p = 0.2713, MMRM — [p-value comment as in outcome 11, analysis 1]; LS Mean Difference = -2.5, 95% CI 2-sided [-7.0 to 2.0], Standard Error of Mean 2.28
Statistical Analysis 3: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 42; Test type: Superiority; p = 0.8048, MMRM — [p-value comment as in outcome 11, analysis 1]; LS Mean Difference = 0.6, 95% CI 2-sided [-4.2 to 5.4], Standard Error of Mean 2.43
Statistical Analysis 4: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 42; Test type: Superiority; p = 0.7665, MMRM — [p-value comment as in outcome 11, analysis 1]; LS Mean Difference = -0.7, 95% CI 2-sided [-5.3 to 3.9], Standard Error of Mean 2.35

12. Secondary Outcome: Change From Baseline in HAM-D Maier Subscale Score
Description: The 17-item HAM-D is used to rate the severity of depression in participants who were already diagnosed as depressed. HAM-D subscale scores are calculated as the sum of the items comprising each subscale. The Maier subscale score is the sum of the following symptom scores, scored in a range of 0 to 4: Depressed mood, feelings of guilt, work and activities, retardation, agitation, and anxiety psychic. Total HAM-D Maier subscale scores were transformed to a scale of 0 to 100. Higher scores indicate more severe depression. A negative change from baseline indicates less depression.
Time Frame: Baseline, Days 15, and 42
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | SAGE-217 Matched Placebo | SAGE-217 20 mg | SAGE-217 30 mg
Number analyzed (Participants) | 141 | 152 | 153
score on a scale
  Change from Baseline at Day 15 | -23.4 (1.34) | -23.1 (1.37) | -25.9 (1.45)
  Change from Baseline at Day 42: number analyzed (Participants) | 135 | 140 | 136
  Change from Baseline at Day 42 | -25.0 (1.42) | -24.8 (1.53) | -26.2 (1.49)
Statistical Analysis 1: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 15; Test type: Superiority; p = 0.8575, MMRM — MMRM with treatment, BL HAM-D Maier subscale score, anti-depressant use at BL, assessment time point, and time point-by-treatment interaction as fixed effects were used for analysis; LS Mean Difference = 0.3, 95% CI 2-sided [-3.4 to 4.1], Standard Error of Mean 1.91
Statistical Analysis 2: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 15; Test type: Superiority; p = 0.1978, MMRM — [p-value comment as in outcome 12, analysis 1]; LS Mean Difference = -2.5, 95% CI 2-sided [-6.3 to 1.3], Standard Error of Mean 1.94
Statistical Analysis 3: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 42; Test type: Superiority; p = 0.9298, MMRM — [p-value comment as in outcome 12, analysis 1]; LS Mean Difference = 0.2, 95% CI 2-sided [-3.9 to 4.3], Standard Error of Mean 2.08
Statistical Analysis 4: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 42; Test type: Superiority; p = 0.5487, MMRM — [p-value comment as in outcome 12, analysis 1]; LS Mean Difference = -1.2, 95% CI 2-sided [-5.2 to 2.8], Standard Error of Mean 2.03

13. Secondary Outcome: Change From Baseline in HAM-D Individual Item Scores
Description: The 17-item HAM-D is used to rate the severity of depression in participants who were already diagnosed as depressed. The HAM-D comprises individual ratings of the following symptoms scored in a range of 0 to 2: Insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight (according to participant), and insight. The following symptoms are scored in a range of 0 to 4: Agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety (psychic and somatic), and hypochondriasis. For each symptom, higher scores indicate more severe depression. A negative change from baseline indicates less depression. A positive change from baseline indicates more depression.
Time Frame: Baseline, Days 15, and 42
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | SAGE-217 Matched Placebo | SAGE-217 20 mg | SAGE-217 30 mg
Number analyzed (Participants) | 141 | 152 | 153
score on a scale
  Depressed Mood: Change from Baseline at Day 15 | -1.3 (0.10) | -1.3 (0.10) | -1.4 (0.10)
  Depressed Mood: Change from Baseline at Day 42: number analyzed (Participants) | 135 | 140 | 136
  Depressed Mood: Change from Baseline at Day 42 | -1.3 (0.10) | -1.3 (0.11) | -1.5 (0.10)
  Feelings of Guilt: Change from Baseline at Day 15 | -1.1 (0.08) | -1.0 (0.07) | -1.1 (0.07)
  Feelings of Guilt: Change from Baseline at Day 42: number analyzed (Participants) | 135 | 140 | 136
  Feelings of Guilt: Change from Baseline at Day 42 | -1.2 (0.08) | -1.1 (0.08) | -1.1 (0.08)
  Suicide: Change from Baseline at Day 15 | -0.3 (0.04) | -0.3 (0.04) | -0.3 (0.04)
  Suicide: Change from Baseline at Day 42: number analyzed (Participants) | 135 | 140 | 136
  Suicide: Change from Baseline at Day 42 | -0.3 (0.04) | -0.3 (0.04) | -0.3 (0.04)
  Insomnia Early - Early Night: Change from Baseline at Day 15 | -0.8 (0.07) | -0.9 (0.07) | -0.8 (0.07)
  Insomnia Early - Early Night: Change from Baseline at Day 42: number analyzed (Participants) | 135 | 140 | 136
  Insomnia Early - Early Night: Change from Baseline at Day 42 | -0.7 (0.07) | -0.6 (0.07) | -0.6 (0.08)
  Insomnia Middle - Middle Night: Change from Baseline at Day 15 | -0.8 (0.06) | -0.9 (0.07) | -0.9 (0.07)
  Insomnia Middle - Middle Night: Change from Baseline at Day 42: number analyzed (Participants) | 135 | 140 | 136
  Insomnia Middle - Middle Night: Change from Baseline at Day 42 | -0.7 (0.07) | -0.7 (0.07) | -0.8 (0.07)
  Insomnia Early Hours - Morning: Change from Baseline at Day 15 | -0.4 (0.06) | -0.5 (0.06) | -0.6 (0.06)
  Insomnia Early Hours - Morning: Change from Baseline at Day 42: number analyzed (Participants) | 135 | 140 | 136
  Insomnia Early Hours - Morning: Change from Baseline at Day 42 | -0.4 (0.07) | -0.4 (0.07) | -0.4 (0.07)
  Work and Activities: Change from Baseline at Day 15 | -1.2 (0.09) | -1.2 (0.10) | -1.3 (0.10)
  Work and Activities: Change from Baseline at Day 42: number analyzed (Participants) | 135 | 140 | 136
  Work and Activities: Change from Baseline at Day 42 | -1.2 (0.10) | -1.3 (0.10) | -1.3 (0.10)
  Retardation: Change from Baseline at Day 15 | -0.5 (0.04) | -0.5 (0.05) | -0.5 (0.05)
  Retardation: Change from Baseline at Day 42: number analyzed (Participants) | 135 | 140 | 136
  Retardation: Change from Baseline at Day 42 | -0.6 (0.04) | -0.5 (0.05) | -0.6 (0.04)
  Agitation: Change from Baseline at Day 15 | -0.5 (0.05) | -0.5 (0.05) | -0.6 (0.05)
  Agitation: Change from Baseline at Day 42: number analyzed (Participants) | 135 | 140 | 136
  Agitation: Change from Baseline at Day 42 | -0.5 (0.05) | -0.6 (0.06) | -0.6 (0.05)
  Anxiety Psychic: Change from Baseline at Day 15 | -1.1 (0.09) | -1.1 (0.09) | -1.4 (0.08)
  Anxiety Psychic: Change from Baseline at Day 42: number analyzed (Participants) | 135 | 140 | 136
  Anxiety Psychic: Change from Baseline at Day 42 | -1.2 (0.09) | -1.2 (0.09) | -1.2 (0.09)
  Anxiety Somatic: Change from Baseline at Day 15 | -0.8 (0.07) | -0.7 (0.06) | -0.8 (0.07)
  Anxiety Somatic: Change from Baseline at Day 42: number analyzed (Participants) | 135 | 140 | 136
  Anxiety Somatic: Change from Baseline at Day 42 | -0.9 (0.08) | -0.8 (0.07) | -0.9 (0.07)
  Somatic Symptoms Gastrointestinal: Change from Baseline at Day 15 | -0.6 (0.06) | -0.6 (0.06) | -0.6 (0.06)
  Somatic Symptoms Gastrointestinal: Change from Baseline at Day 42: number analyzed (Participants) | 135 | 140 | 136
  Somatic Symptoms Gastrointestinal: Change from Baseline at Day 42 | -0.6 (0.06) | -0.7 (0.07) | -0.7 (0.06)
  General Somatic Symptoms: Change from Baseline at Day 15 | -0.6 (0.06) | -0.7 (0.06) | -0.7 (0.06)
  General Somatic Symptoms: Change from Baseline at Day 42: number analyzed (Participants) | 135 | 140 | 136
  General Somatic Symptoms: Change from Baseline at Day 42 | -0.6 (0.07) | -0.6 (0.07) | -0.7 (0.07)
  Genital Symptoms: Change from Baseline at Day 15 | -0.5 (0.07) | -0.5 (0.06) | -0.6 (0.07)
  Genital Symptoms: Change from Baseline at Day 42: number analyzed (Participants) | 135 | 140 | 136
  Genital Symptoms: Change from Baseline at Day 42 | -0.5 (0.07) | -0.5 (0.07) | -0.6 (0.07)
  Hypochondriasis: Change from Baseline at Day 15 | -0.4 (0.05) | -0.4 (0.05) | -0.5 (0.05)
  Hypochondriasis: Change from Baseline at Day 42: number analyzed (Participants) | 135 | 140 | 136
  Hypochondriasis: Change from Baseline at Day 42 | -0.6 (0.04) | -0.5 (0.05) | -0.5 (0.05)
  Loss of Weight: Change from Baseline at Day 15 | -0.4 (0.05) | -0.4 (0.05) | -0.4 (0.06)
  Loss of Weight: Change from Baseline at Day 42: number analyzed (Participants) | 135 | 140 | 136
  Loss of Weight: Change from Baseline at Day 42 | -0.4 (0.06) | -0.4 (0.05) | -0.4 (0.06)
  Insight: Change from Baseline at Day 15 | 0.0 (0.02) | 0.0 (0.02) | -0.1 (0.01)
  Insight: Change from Baseline at Day 42: number analyzed (Participants) | 135 | 140 | 136
  Insight: Change from Baseline at Day 42 | 0.0 (0.02) | 0.0 (0.01) | 0.0 (0.02)
Statistical Analysis 1: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 15: Depressed Mood; Test type: Superiority; p = 0.6270, MMRM — MMRM with treatment, each BL individual item HAM-D score, anti-depressant use at BL, assessment time point, and time point-by-treatment interaction as fixed effects were used for analysis; LS Mean Difference = 0.1, 95% CI 2-sided [-0.2 to 0.3], Standard Error of Mean 0.14
Statistical Analysis 2: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 15: Depressed Mood; Test type: Superiority; p = 0.5463, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.4 to 0.2], Standard Error of Mean 0.14
Statistical Analysis 3: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 42: Depressed Mood; Test type: Superiority; p = 0.8716, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.3 to 0.3], Standard Error of Mean 0.15
Statistical Analysis 4: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 42: Depressed Mood; Test type: Superiority; p = 0.4383, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.4 to 0.2], Standard Error of Mean 0.14
Statistical Analysis 5: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 15: Feelings of Guilt; Test type: Superiority; p = 0.4794, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.1, 95% CI 2-sided [-0.1 to 0.3], Standard Error of Mean 0.10
Statistical Analysis 6: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 15: Feelings of Guilt; Test type: Superiority; p = 0.9717, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.2 to 0.2], Standard Error of Mean 0.10
Statistical Analysis 7: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 42: Feelings of Guilt; Test type: Superiority; p = 0.3701, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.1, 95% CI 2-sided [-0.1 to 0.3], Standard Error of Mean 0.11
Statistical Analysis 8: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 42: Feelings of Guilt; Test type: Superiority; p = 0.3972, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.1, 95% CI 2-sided [-0.1 to 0.3], Standard Error of Mean 0.11
Statistical Analysis 9: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 15: Suicide; Test type: Superiority; p = 0.5761, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.1 to 0.1], Standard Error of Mean 0.06
Statistical Analysis 10: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 15: Suicide; Test type: Superiority; p = 0.4379, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.1 to 0.1], Standard Error of Mean 0.05
Statistical Analysis 11: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 42: Suicide; Test type: Superiority; p = 0.6087, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.1 to 0.1], Standard Error of Mean 0.06
Statistical Analysis 12: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 42: Suicide; Test type: Superiority; p = 0.9791, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.1 to 0.1], Standard Error of Mean 0.05
Statistical Analysis 13: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 15: Insomnia Early - Early Night; Test type: Superiority; p = 0.2093, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.3 to 0.1], Standard Error of Mean 0.10
Statistical Analysis 14: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 15: Insomnia Early - Early Night; Test type: Superiority; p = 0.5189, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.3 to 0.1], Standard Error of Mean 0.10
Statistical Analysis 15: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 42: Insomnia Early - Early Night; Test type: Superiority; p = 0.6617, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.2 to 0.2], Standard Error of Mean 0.10
Statistical Analysis 16: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 42: Insomnia Early - Early Night; Test type: Superiority; p = 0.2632, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.1, 95% CI 2-sided [-0.1 to 0.3], Standard Error of Mean 0.10
Statistical Analysis 17: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 15: Insomnia Middle - Middle Night; Test type: Superiority; p = 0.2740, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.3 to 0.1], Standard Error of Mean 0.09
Statistical Analysis 18: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 15: Insomnia Middle - Middle Night; Test type: Superiority; p = 0.1185, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.3 to 0.0], Standard Error of Mean 0.09
Statistical Analysis 19: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 42: Insomnia Middle - Middle Night; Test type: Superiority; p = 0.9450, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.2 to 0.2], Standard Error of Mean 0.10
Statistical Analysis 20: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 42: Insomnia Middle - Middle Night; Test type: Superiority; p = 0.6343, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.2 to 0.1], Standard Error of Mean 0.09
Statistical Analysis 21: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 15: Insomnia Early Hours - Morning; Test type: Superiority; p = 0.3169, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.3 to 0.1], Standard Error of Mean 0.09
Statistical Analysis 22: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 15: Insomnia Early Hours - Morning; Test type: Superiority; p = 0.0178, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -0.2, 95% CI 2-sided [-0.4 to 0.0], Standard Error of Mean 0.09
Statistical Analysis 23: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 42: Insomnia Early Hours - Morning; Test type: Superiority; p = 0.8504, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.2 to 0.2], Standard Error of Mean 0.10
Statistical Analysis 24: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 42: Insomnia Early Hours - Morning; Test type: Superiority; p = 0.5647, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.2 to 0.1], Standard Error of Mean 0.10
Statistical Analysis 25: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 15: Work and Activities; Test type: Superiority; p = 0.5914, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.3 to 0.2], Standard Error of Mean 0.14
Statistical Analysis 26: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 15: Work and Activities; Test type: Superiority; p = 0.4603, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.4 to 0.2], Standard Error of Mean 0.14
Statistical Analysis 27: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 42: Work and Activities; Test type: Superiority; p = 0.5637, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.4 to 0.2], Standard Error of Mean 0.15
Statistical Analysis 28: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 42: Work and Activities; Test type: Superiority; p = 0.4638, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.4 to 0.2], Standard Error of Mean 0.14
Statistical Analysis 29: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 15: Retardation; Test type: Superiority; p = 0.1846, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.1, 95% CI 2-sided [0.0 to 0.2], Standard Error of Mean 0.07
Statistical Analysis 30: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 15: Retardation; Test type: Superiority; p = 0.4837, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.1 to 0.2], Standard Error of Mean 0.06
Statistical Analysis 31: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 42: Retardation; Test type: Superiority; p = 0.1178, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.1, 95% CI 2-sided [0.0 to 0.2], Standard Error of Mean 0.07
Statistical Analysis 32: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 42: Retardation; Test type: Superiority; p = 0.7888, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.1 to 0.1], Standard Error of Mean 0.06
Statistical Analysis 33: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 15: Agitation; Test type: Superiority; p = 0.9496, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.1 to 0.1], Standard Error of Mean 0.07
Statistical Analysis 34: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 15: Agitation; Test type: Superiority; p = 0.0497, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.3 to 0.0], Standard Error of Mean 0.07
Statistical Analysis 35: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 42: Agitation; Test type: Superiority; p = 0.4189, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.2 to 0.1], Standard Error of Mean 0.08
Statistical Analysis 36: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 42: Agitation; Test type: Superiority; p = 0.1342, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.3 to 0.0], Standard Error of Mean 0.08
Statistical Analysis 37: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 15: Anxiety Psychic; Test type: Superiority; p = 0.9202, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.3 to 0.2], Standard Error of Mean 0.12
Statistical Analysis 38: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 15: Anxiety Psychic; Test type: Superiority; p = 0.0260, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -0.3, 95% CI 2-sided [-0.5 to 0.0], Standard Error of Mean 0.12
Statistical Analysis 39: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 42: Anxiety Psychic; Test type: Superiority; p = 0.9370, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.3 to 0.2], Standard Error of Mean 0.13
Statistical Analysis 40: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 42: Anxiety Psychic; Test type: Superiority; p = 0.8440, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.3 to 0.2], Standard Error of Mean 0.13
Statistical Analysis 41: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 15: Anxiety Somatic; Test type: Superiority; p = 0.4480, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.1, 95% CI 2-sided [-0.1 to 0.3], Standard Error of Mean 0.09
Statistical Analysis 42: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 15: Anxiety Somatic; Test type: Superiority; p = 0.6345, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.1 to 0.2], Standard Error of Mean 0.09
Statistical Analysis 43: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 42: Anxiety Somatic; Test type: Superiority; p = 0.4123, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.1, 95% CI 2-sided [-0.1 to 0.3], Standard Error of Mean 0.10
Statistical Analysis 44: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 42: Anxiety Somatic; Test type: Superiority; p = 0.7523, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.2 to 0.2], Standard Error of Mean 0.10
Statistical Analysis 45: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 15: Somatic Symptoms Gastrointestinal; Test type: Superiority; p = 0.6505, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.2 to 0.1], Standard Error of Mean 0.09
Statistical Analysis 46: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 15: Somatic Symptoms Gastrointestinal; Test type: Superiority; p = 0.3674, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.3 to 0.1], Standard Error of Mean 0.09
Statistical Analysis 47: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 42: Somatic Symptoms Gastrointestinal; Test type: Superiority; p = 0.8360, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.2 to 0.2], Standard Error of Mean 0.09
Statistical Analysis 48: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 42: Somatic Symptoms Gastrointestinal; Test type: Superiority; p = 0.6870, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.2 to 0.1], Standard Error of Mean 0.09
Statistical Analysis 49: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 15: General Somatic Symptoms; Test type: Superiority; p = 0.1364, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.3 to 0.0], Standard Error of Mean 0.08
Statistical Analysis 50: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 15: General Somatic Symptoms; Test type: Superiority; p = 0.1578, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.3 to 0.0], Standard Error of Mean 0.09
Statistical Analysis 51: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 42: General Somatic Symptoms; Test type: Superiority; p = 0.9062, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.2 to 0.2], Standard Error of Mean 0.09
Statistical Analysis 52: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 42: General Somatic Symptoms; Test type: Superiority; p = 0.8596, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.2 to 0.2], Standard Error of Mean 0.09
Statistical Analysis 53: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 15: Genital Symptoms; Test type: Superiority; p = 0.9488, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.2 to 0.2], Standard Error of Mean 0.09
Statistical Analysis 54: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 15: Genital Symptoms; Test type: Superiority; p = 0.1514, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.3 to 0.0], Standard Error of Mean 0.09
Statistical Analysis 55: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 42: Genital Symptoms; Test type: Superiority; p = 0.5796, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.2 to 0.1], Standard Error of Mean 0.09
Statistical Analysis 56: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 42: Genital Symptoms; Test type: Superiority; p = 0.4739, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.3 to 0.1], Standard Error of Mean 0.10
Statistical Analysis 57: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 15: Hypochondriasis; Test type: Superiority; p = 0.9439, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.1 to 0.1], Standard Error of Mean 0.07
Statistical Analysis 58: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 15: Hypochondriasis; Test type: Superiority; p = 0.3891, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.2 to 0.1], Standard Error of Mean 0.07
Statistical Analysis 59: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 42: Hypochondriasis; Test type: Superiority; p = 0.0308, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.1, 95% CI 2-sided [0.0 to 0.3], Standard Error of Mean 0.07
Statistical Analysis 60: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 42: Hypochondriasis; Test type: Superiority; p = 0.0620, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.1, 95% CI 2-sided [0.0 to 0.3], Standard Error of Mean 0.07
Statistical Analysis 61: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 15: Loss of Weight; Test type: Superiority; p = 0.7744, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.2 to 0.1], Standard Error of Mean 0.07
Statistical Analysis 62: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 15: Loss of Weight; Test type: Superiority; p = 0.9312, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.1 to 0.2], Standard Error of Mean 0.08
Statistical Analysis 63: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 42: Loss of Weight; Test type: Superiority; p = 0.3105, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.2 to 0.1], Standard Error of Mean 0.08
Statistical Analysis 64: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 42: Loss of Weight; Test type: Superiority; p = 0.8406, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.1 to 0.2], Standard Error of Mean 0.08
Statistical Analysis 65: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 15: Insight; Test type: Superiority; p = 0.4834, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.1 to 0.0], Standard Error of Mean 0.03
Statistical Analysis 66: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 15: Insight; Test type: Superiority; p = 0.0961, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.1 to 0.0], Standard Error of Mean 0.02
Statistical Analysis 67: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 42: Insight; Test type: Superiority; p = 0.8290, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [0.0 to 0.0], Standard Error of Mean 0.02
Statistical Analysis 68: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 42: Insight; Test type: Superiority; p = 0.9546, MMRM — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [0.0 to 0.0], Standard Error of Mean 0.02

14. Secondary Outcome: Change From Baseline in Insomnia Severity Index (ISI) Total Score
Description: The ISI is a validated questionnaire designed to assess the nature, severity, and impact of insomnia. The ISI uses a 5-point Likert scale to measure various aspects of insomnia severity (0=none, 1=mild, 2=moderate; 3=severe; 4=very severe), satisfaction with current sleep pattern (0=very satisfied, 1=satisfied, 2=moderately satisfied, 3=dissatisfied, 4=very dissatisfied), and various aspects of the impact of insomnia on daily functioning (0=not at all, 1=a little, 2=somewhat, 3=much, 4=very much). The ISI total score is calculated as the sum of the 7 individual item scores and the possible total score range is from 0 to 28, categorized as follows: 0 to 7=no clinically significant insomnia, 8 to 14=subthreshold insomnia, 15 to 21=clinical insomnia (moderate severity), and 22 to 28=clinical insomnia (severe). Higher scores indicate more severity. A negative change from baseline indicates less severe insomnia.
Time Frame: Baseline, Days 15, and 42
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | SAGE-217 Matched Placebo | SAGE-217 20 mg | SAGE-217 30 mg
Number analyzed (Participants) | 141 | 152 | 153
score on a scale
  Change from Baseline at Day 15 | -6.2 (0.55) | -7.4 (0.58) | -8.2 (0.58)
  Change from Baseline at Day 42: number analyzed (Participants) | 135 | 141 | 137
  Change from Baseline at Day 42 | -6.9 (0.64) | -5.9 (0.60) | -6.9 (0.62)
Statistical Analysis 1: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 15; Test type: Superiority; p = 0.1308, MMRM — MMRM with treatment, BL ISI total score, anti-depressant use at BL, assessment time point, and time point-by-treatment interaction as fixed effects were used for analysis; LS Mean Difference = -1.2, 95% CI 2-sided [-2.7 to 0.4], Standard Error of Mean 0.78
Statistical Analysis 2: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 15; Test type: Superiority; p = 0.0096, MMRM — [p-value comment as in outcome 14, analysis 1]; LS Mean Difference = -2.0, 95% CI 2-sided [-3.5 to -0.5], Standard Error of Mean 0.77
Statistical Analysis 3: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 42; Test type: Superiority; p = 0.2674, MMRM — [p-value comment as in outcome 14, analysis 1]; LS Mean Difference = 1.0, 95% CI 2-sided [-0.7 to 2.7], Standard Error of Mean 0.86
Statistical Analysis 4: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 42; Test type: Superiority; p = 0.9771, MMRM — [p-value comment as in outcome 14, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-1.7 to 1.7], Standard Error of Mean 0.87

15. Secondary Outcome: Change From Baseline in Core Consensus Sleep Diary Parameters: Sleep Onset Latency (sSL), Wake After Sleep Onset (sWASO), and Total Sleep Time (sTST)
Description: The Core Consensus Sleep Diary collected subjective responses to a series of questions related to participant's daily sleep pattern (i.e., time to bed, time to fall asleep, time to final awakening, and a question related to quality of sleep) to derive sleep parameters, including sSL, sTST, and sWASO. The take-home participant sleep diary assessment was administered using an eDiary solution. The eDiary was captured using either a provisioned smartphone device or a bring-your-own-device solution, depending on the participant's preference. sTST is a derived parameter calculated as: Time of final awakening - (time when tried to sleep + time taken to fall asleep)-time of being awake after sleep onset. Negative change from baseline in sSL and sWASO indicates improvement. Positive change from baseline in sTST indicates improvement.
Time Frame: Baseline, Days 15, and 28
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | SAGE-217 Matched Placebo | SAGE-217 20 mg | SAGE-217 30 mg
Number analyzed (Participants) | 129 | 138 | 143
minutes
  Change from Baseline in sSL at Day 15 | -12.2 (3.02) | -14.4 (3.34) | -20.1 (3.24)
  Change from Baseline in sSL at Day 28: number analyzed (Participants) | 92 | 114 | 94
  Change from Baseline in sSL at Day 28 | -12.1 (4.26) | -16.4 (3.73) | -15.8 (4.77)
  Change from Baseline in sWASO at Day 15 | -19.2 (2.87) | -21.4 (3.00) | -18.8 (4.28)
  Change from Baseline in sWASO at Day 28: number analyzed (Participants) | 92 | 114 | 94
  Change from Baseline in sWASO at Day 28 | -21.0 (3.68) | -18.2 (3.18) | -17.1 (4.57)
  Change from Baseline in sTST at Day 15: number analyzed (Participants) | 124 | 135 | 138
  Change from Baseline in sTST at Day 15 | 30.1 (7.92) | 54.2 (7.36) | 47.5 (7.99)
  Change from Baseline in sTST at Day 28: number analyzed (Participants) | 88 | 112 | 91
  Change from Baseline in sTST at Day 28 | 27.1 (9.93) | 41.2 (10.41) | 37.4 (9.36)
Statistical Analysis 1: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 15: sSL; Test type: Superiority; p = 0.6110, MMRM — MMRM with treatment, BL sSL score, anti-depressant use at BL, assessment time point, and time point-by-treatment interaction as fixed effects were used for analysis; LS Mean Difference = -2.2, 95% CI 2-sided [-10.9 to 6.4], Standard Error of Mean 4.42
Statistical Analysis 2: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 15: sSL; Test type: Superiority; p = 0.0581, MMRM — [p-value comment as in outcome 15, analysis 1]; LS Mean Difference = -8.0, 95% CI 2-sided [-16.2 to 0.3], Standard Error of Mean 4.19
Statistical Analysis 3: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 28: sSL; Test type: Superiority; p = 0.4493, MMRM — [p-value comment as in outcome 15, analysis 1]; LS Mean Difference = -4.3, 95% CI 2-sided [-15.5 to 6.9], Standard Error of Mean 5.68
Statistical Analysis 4: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 28: sSL; Test type: Superiority; p = 0.5587, MMRM — [p-value comment as in outcome 15, analysis 1]; LS Mean Difference = -3.7, 95% CI 2-sided [-16.0 to 8.6], Standard Error of Mean 6.25
Statistical Analysis 5: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 15: sWASO; Test type: Superiority; p = 0.5976, MMRM — MMRM with treatment, BL sWASO score, anti-depressant use at BL, assessment time point, and time point-by-treatment interaction as fixed effects were used for analysis; LS Mean Difference = -2.1, 95% CI 2-sided [-10.1 to 5.8], Standard Error of Mean 4.06
Statistical Analysis 6: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 15: sWASO; Test type: Superiority; p = 0.9421, MMRM — [p-value comment as in outcome 15, analysis 5]; LS Mean Difference = 0.4, 95% CI 2-sided [-9.6 to 10.3], Standard Error of Mean 5.05
Statistical Analysis 7: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 28: sWASO; Test type: Superiority; p = 0.5581, MMRM — [p-value comment as in outcome 15, analysis 5]; LS Mean Difference = 2.9, 95% CI 2-sided [-6.7 to 12.4], Standard Error of Mean 4.86
Statistical Analysis 8: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 28: sWASO; Test type: Superiority; p = 0.4997, MMRM — [p-value comment as in outcome 15, analysis 5]; LS Mean Difference = 3.9, 95% CI 2-sided [-7.5 to 15.4], Standard Error of Mean 5.82
Statistical Analysis 9: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 15: sTST; Test type: Superiority; p = 0.0224, MMRM — MMRM with treatment, BL sTST score, anti-depressant use at BL, assessment time point, and time point-by-treatment interaction as fixed effects were used for analysis; LS Mean Difference = 24.0, 95% CI 2-sided [3.4 to 44.7], Standard Error of Mean 10.50
Statistical Analysis 10: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 15: sTST; Test type: Superiority; p = 0.1117, MMRM — [p-value comment as in outcome 15, analysis 9]; LS Mean Difference = 17.4, 95% CI 2-sided [-4.1 to 38.9], Standard Error of Mean 10.93
Statistical Analysis 11: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 28: sTST; Test type: Superiority; p = 0.3208, MMRM — [p-value comment as in outcome 15, analysis 9]; LS Mean Difference = 14.1, 95% CI 2-sided [-13.8 to 42.0], Standard Error of Mean 14.18
Statistical Analysis 12: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 28: sTST; Test type: Superiority; p = 0.4440, MMRM — [p-value comment as in outcome 15, analysis 9]; LS Mean Difference = 10.3, 95% CI 2-sided [-16.1 to 36.6], Standard Error of Mean 13.40

16. Secondary Outcome: Change From Baseline in Core Consensus Sleep Diary Parameter: Number of Awakenings (sNAW)
Description: The Core Consensus Sleep Diary was used to collect subjective sleep parameter of sNAW. sNAW was calculated from the onset of persistent sleep until lights on. An awakening is defined as at least 2 consecutive epochs of wake. Individual awakenings were separated by at least 1 epoch of Stage N2 (also fairly light, with sudden increases in brain wave frequency known as sleep spindles), N3 (slow wave or deep sleep) or rapid eye movement (REM) sleep. Lower ratings indicate better sleep quality and more refreshing/restorative quality of sleep.
Time Frame: Baseline, Days 15, and 28
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: awakenings
Arm/Group | SAGE-217 Matched Placebo | SAGE-217 20 mg | SAGE-217 30 mg
Number analyzed (Participants) | 129 | 138 | 143
awakenings
  Change from Baseline at Day 15 | -0.4 (0.07) | -0.5 (0.07) | -0.7 (0.07)
  Change from Baseline at Day 28: number analyzed (Participants) | 92 | 114 | 94
  Change from Baseline at Day 28 | -0.5 (0.08) | -0.3 (0.09) | -0.5 (0.09)
Statistical Analysis 1: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 15; Test type: Superiority; p = 0.4737, MMRM — MMRM with treatment, BL sNAW score, anti-depressant use at BL, assessment time point, and time point-by-treatment interaction as fixed effects were used for analysis; LS Mean Difference = -0.1, 95% CI 2-sided [-0.3 to 0.1], Standard Error of Mean 0.10
Statistical Analysis 2: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 15; Test type: Superiority; p = 0.0138, MMRM — [p-value comment as in outcome 16, analysis 1]; LS Mean Difference = -0.2, 95% CI 2-sided [-0.4 to 0.0], Standard Error of Mean 0.10
Statistical Analysis 3: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 28; Test type: Superiority; p = 0.1098, MMRM — [p-value comment as in outcome 16, analysis 1]; LS Mean Difference = 0.2, 95% CI 2-sided [0.0 to 0.4], Standard Error of Mean 0.12
Statistical Analysis 4: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 28; Test type: Superiority; p = 0.6234, MMRM — [p-value comment as in outcome 16, analysis 1]; LS Mean Difference = 0.1, 95% CI 2-sided [-0.2 to 0.3], Standard Error of Mean 0.11

17. Secondary Outcome: Change From Baseline in Core Consensus Sleep Diary Parameter: Number of Participants With Subjective Sleep Quality (sSQ) Response
Description: The Core Consensus Sleep Diary collected subjective sleep parameters, including sleep quality (sSQ). The take-home participant sleep diary assessment was administered using an eDiary solution. The eDiary was captured using either a provisioned smartphone device or a bring-your-own-device solution, depending on the participant's preference. sSQ is rated on a 5-point Likert scale ranging from 1 (very poor) to 5 (very good). Higher ratings indicate better sleep quality. sSQ response is defined as having a sSQ score of very good or good.
Time Frame: Baseline, Days 15, and 28
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | SAGE-217 Matched Placebo | SAGE-217 20 mg | SAGE-217 30 mg
Number analyzed (Participants) | 132 | 143 | 146
Participants
  Change from Baseline at Day 15 | 36 | 35 | 32
  Change from Baseline at Day 28: number analyzed (Participants) | 94 | 117 | 96
  Change from Baseline at Day 28 | 30 | 35 | 28
Statistical Analysis 1: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 15; Test type: Superiority; p = 0.6741, GEE — GEE for binary response model, with factors for treatment, BL sleep quality response, anti-depressant use at BL, assessment time point, and time point-by-treatment interaction were used for analysis; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.52 to 1.53]
Statistical Analysis 2: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 15; Test type: Superiority; p = 0.3924, GEE — [p-value comment as in outcome 17, analysis 1]; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.46 to 1.36]
Statistical Analysis 3: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 28; Test type: Superiority; p = 0.7307, GEE — [p-value comment as in outcome 17, analysis 1]; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.51 to 1.60]
Statistical Analysis 4: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 28; Test type: Superiority; p = 0.8358, GEE — [p-value comment as in outcome 17, analysis 1]; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.52 to 1.70]

18. Secondary Outcome: Change From Baseline in the 36-item Short Form Survey Version 2 (SF-36v2) Physical and Mental Component Summary Scores
Description: Participant's health was assessed using Patient-reported outcome (PRO) health related quality of life (HRQOL), SF-36v2 which is a 36-item measure of health status. It covers eight health dimensions including four physical health status domains (physical functioning, role participation with physical health problems, bodily pain, and general health) and four mental health status domains (vitality, social functioning, role participation with emotional health problems, and mental health). Two summary scores, physical component summary (PCS), and mental component summary (MCS) were produced by taking a weighted linear combination of the eight individual domains. The score range for PCS and MCS is 0 to 100 (100=highest level of functioning). Higher scores indicate a better state of health. A negative change from baseline indicates deteriorating health.
Time Frame: Baseline, Days 15, and 42
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | SAGE-217 Matched Placebo | SAGE-217 20 mg | SAGE-217 30 mg
Number analyzed (Participants) | 140 | 152 | 153
score on a scale
  PCS Score: Change from Baseline at Day 15 | -0.9 (0.56) | -1.2 (0.48) | -1.4 (0.52)
  PCS Score: Change from Baseline at Day 42: number analyzed (Participants) | 135 | 140 | 137
  PCS Score: Change from Baseline at Day 42 | -1.9 (0.63) | -2.1 (0.50) | -1.3 (0.58)
  MCS Score: Change from Baseline at Day 15 | 13.4 (1.15) | 14.6 (1.20) | 16.0 (1.31)
  MCS Score: Change from Baseline at Day 42: number analyzed (Participants) | 135 | 140 | 137
  MCS Score: Change from Baseline at Day 42 | 15.4 (1.21) | 15.9 (1.28) | 16.9 (1.30)
Statistical Analysis 1: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 15: PCS Score; Test type: Superiority; p = 0.7375, MMRM — MMRM with treatment, BL SF-36v2 physical component score, anti-depressant use at BL, assessment time point, and time point-by-treatment interaction as fixed effects were used for analysis; LS Mean Difference = -0.2, 95% CI 2-sided [-1.6 to 1.2], Standard Error of Mean 0.72
Statistical Analysis 2: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 15: PCS Score; Test type: Superiority; p = 0.5144, MMRM — [p-value comment as in outcome 18, analysis 1]; LS Mean Difference = -0.5, 95% CI 2-sided [-1.9 to 1.0], Standard Error of Mean 0.74
Statistical Analysis 3: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 42: PCS Score; Test type: Superiority; p = 0.8343, MMRM — [p-value comment as in outcome 18, analysis 1]; LS Mean Difference = -0.2, 95% CI 2-sided [-1.7 to 1.4], Standard Error of Mean 0.79
Statistical Analysis 4: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 42: PCS Score; Test type: Superiority; p = 0.4569, MMRM — [p-value comment as in outcome 18, analysis 1]; LS Mean Difference = 0.6, 95% CI 2-sided [-1.0 to 2.3], Standard Error of Mean 0.85
Statistical Analysis 5: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 15: MCS Score; Test type: Superiority; p = 0.4663, MMRM — MMRM with treatment, BL SF-36v2 mental component score, anti-depressant use at BL, assessment time point, and time point-by-treatment interaction as fixed effects were used for analysis; LS Mean Difference = 1.2, 95% CI 2-sided [-2.0 to 4.4], Standard Error of Mean 1.63
Statistical Analysis 6: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 15: MCS Score; Test type: Superiority; p = 0.1138, MMRM — [p-value comment as in outcome 18, analysis 5]; LS Mean Difference = 2.7, 95% CI 2-sided [-0.6 to 6.0], Standard Error of Mean 1.68
Statistical Analysis 7: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 42: MCS Score; Test type: Superiority; p = 0.7901, MMRM — [p-value comment as in outcome 18, analysis 5]; LS Mean Difference = 0.5, 95% CI 2-sided [-3.0 to 3.9], Standard Error of Mean 1.74
Statistical Analysis 8: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 42: MCS Score; Test type: Superiority; p = 0.3955, MMRM — [p-value comment as in outcome 18, analysis 5]; LS Mean Difference = 1.5, 95% CI 2-sided [-1.9 to 4.8], Standard Error of Mean 1.71

19. Secondary Outcome: Change From Baseline in the 9-item Patient Health Questionnaire (PHQ-9) Total Score
Description: The PHQ-9 is a participant-rated depressive symptom severity scale to monitor severity over time for newly diagnosed participants or participants in current treatment for depression. Scoring was based on participants' responses to each of the 9 questions, as follows: 0=not at all; 1=several days; 2=more than half the days; and 3=nearly every day. The PHQ-9 total score was calculated as the sum of the 9 individual item scores. The PHQ-9 total score was categorized as follows: 1 to 4=minimal depression, 5 to 9=mild depression, 10 to 14=moderate depression, 15 to 19=moderately severe depression; and 20 to 27=severe depression. Higher scores indicate more severe depression. A negative change from baseline indicates reduced depression.
Time Frame: Baseline, Days 15, and 42
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | SAGE-217 Matched Placebo | SAGE-217 20 mg | SAGE-217 30 mg
Number analyzed (Participants) | 139 | 152 | 149
score on a scale
  Change from Baseline at Day 15 | -7.1 (0.59) | -7.3 (0.60) | -8.3 (0.62)
  Change from Baseline at Day 42: number analyzed (Participants) | 135 | 139 | 132
  Change from Baseline at Day 42 | -8.1 (0.61) | -7.3 (0.59) | -8.7 (0.60)
Statistical Analysis 1: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 15; Test type: Superiority; p = 0.8821, MMRM — MMRM with treatment, BL PHQ-9 total score, anti-depressant use at BL, assessment time point, and time point-by-treatment interaction were used for analysis; LS Mean Difference = -0.1, 95% CI 2-sided [-1.8 to 1.5], Standard Error of Mean 0.83
Statistical Analysis 2: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 15; Test type: Superiority; p = 0.1510, MMRM — [p-value comment as in outcome 19, analysis 1]; LS Mean Difference = -1.2, 95% CI 2-sided [-2.8 to 0.4], Standard Error of Mean 0.83
Statistical Analysis 3: Comparison: SAGE-217 Matched Placebo vs SAGE-217 20 mg; Day 42; Test type: Superiority; p = 0.2926, MMRM — [p-value comment as in outcome 19, analysis 1]; LS Mean Difference = 0.9, 95% CI 2-sided [-0.8 to 2.5], Standard Error of Mean 0.84
Statistical Analysis 4: Comparison: SAGE-217 Matched Placebo vs SAGE-217 30 mg; Day 42; Test type: Superiority; p = 0.4785, MMRM — [p-value comment as in outcome 19, analysis 1]; LS Mean Difference = -0.6, 95% CI 2-sided [-2.2 to 1.0], Standard Error of Mean 0.83

20. Secondary Outcome: Number of Participants Who Experienced at Least One Treatment-emergent Adverse Event (TEAE) and Serious TEAE in Treatment and FU Periods
Description: An adverse event (AE) is any untoward medical occurrence in a participant administered with a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of an IP whether or not related to the product. An AE can include any undesirable medical condition, even if no study treatment has been administered. A TEAE is defined as an AE with onset after the start of IP, or any worsening of a pre-existing medical condition/AE with onset after the start of IP and throughout the study. A serious TEAE is defined as a TEAE that at any dose results in death, is immediately life-threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability or incapacity, or results in a congenital abnormality or birth defect.
Time Frame: Treatment period: Up to Day 14; FU period: Day 15 to 42
Population: Safety Set included all participants who were administered IP in treatment period. The AE data were collected and reported period-wise.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment Period: SAGE-217 Matched Placebo: Participants self-administered SAGE-217 matched placebo capsules, orally, once daily in the evening with food for 14 days.
- Treatment Period: SAGE-217 20 mg: Participants self-administered SAGE-217 20 mg capsules, orally, once daily in the evening with food for 14 days.
- Treatment Period: SAGE-217 30 mg: Participants self-administered SAGE-217 30 mg capsules, orally, once daily in the evening with food for 14 days.
- FU Period: SAGE-217 Matched Placebo: Participants who received SAGE-217 matched placebo during the treatment period were included in this group and followed up for 28 days.
- FU Period: SAGE-217 20 mg: Participants who received SAGE-217 20 mg during the treatment period were included in this group and followed up for 28 days.
- FU Period: SAGE-217 30 mg: Participants who received SAGE-217 30 mg during the treatment period were included in this group and followed up for 28 days.
Arm/Group | Treatment Period: SAGE-217 Matched Placebo | Treatment Period: SAGE-217 20 mg | Treatment Period: SAGE-217 30 mg | FU Period: SAGE-217 Matched Placebo | FU Period: SAGE-217 20 mg | FU Period: SAGE-217 30 mg
Number analyzed (Participants) | 190 | 188 | 192 | 190 | 188 | 192
Participants
  TEAE | 77 | 78 | 93 | 46 | 44 | 46
  Serious TEAE | 0 | 0 | 2 | 1 | 1 | 1

21. Secondary Outcome: Number of Participants Who Experienced at Least One Treatment-emergent Adverse Event (TEAE) and Serious TEAE in Extended FU Period
Description: as for outcome 20
Time Frame: Extended FU Period: Day 43 to 182
Population: Extended FU Safety Set included all participants in the Safety Set of treatment period who consented or reconsented to participate in the study in the 6-month FU Period. The AE data were collected and reported period-wise.
Measure: Count of Participants; unit: Participants
Groups:
- Extended FU Period: SAGE-217 Matched Placebo: Participants who received SAGE-217 matched placebo during the treatment period were followed up through Day 182 (6 months following the last IP dose) as a part of the extended FU period.
- Extended FU Period: SAGE-217 20 mg: Participants who received SAGE-217 20 mg during the treatment period were followed up through Day 182 (6 months following the last IP dose) as a part of the extended FU period.
- Extended FU Period: SAGE-217 30 mg: Participants who received SAGE-217 30 mg during the treatment period were followed up through Day 182 (6 months following the last IP dose) as a part of the extended FU period.
Arm/Group | Extended FU Period: SAGE-217 Matched Placebo | Extended FU Period: SAGE-217 20 mg | Extended FU Period: SAGE-217 30 mg
Number analyzed (Participants) | 129 | 127 | 131
Participants
  TEAE | 27 | 29 | 28
  Serious TEAE | 1 | 3 | 1

22. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Laboratory Measures in Treatment and FU Periods
Description: Laboratory parameters include serum chemistry- Alanine aminotransferase: >3x upper limit of normal (ULN); Alanine aminotransferase or aspartate aminotransferase: >3x ULN; Bilirubin: >1.5x ULN, >2x ULN; Calcium: <2.0 millimoles per liter (mmol/L); Gamma Glutamyl Transferase [units per liter (U/L)]: >3xULN; Potassium: >5.4 mmol/L; Sodium: >150 mmol/L; Hematology- Hematocrit : Male <0.385 liter/liter (L/L) and Female <0.345 L/L and Male >0.55 L/L and Female >0.49 L/L; Hemoglobin: Male <115 grams/liter (g/L) and Female <100 g/L; Neutrophils: <1.5 10^9/L.
Time Frame: Treatment period: Up to Day 14; FU period: Day 15 to 42
Population: Safety Set included all participants who were administered IP in treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period: SAGE-217 Matched Placebo | Treatment Period: SAGE-217 20 mg | Treatment Period: SAGE-217 30 mg | FU Period: SAGE-217 Matched Placebo | FU Period: SAGE-217 20 mg | FU Period: SAGE-217 30 mg
Number analyzed (Participants) | 190 | 188 | 192 | 190 | 188 | 192
Participants | 0 | 0 | 0 | 0 | 0 | 0

23. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Laboratory Measures in Extended FU Period
Description: as for outcome 22
Time Frame: Extended FU Period: Day 43 to 182
Population: Extended FU Safety Set included all participants in the Safety Set of treatment period who consented or reconsented to participate in the study in the 6-month FU period.
Measure: Count of Participants; unit: Participants
Arm/Group | Extended FU Period: SAGE-217 Matched Placebo | Extended FU Period: SAGE-217 20 mg | Extended FU Period: SAGE-217 30 mg
Number analyzed (Participants) | 129 | 127 | 131
Participants | 0 | 0 | 0

24. Secondary Outcome: Number of Participants With Clinically Significant Vital Sign Abnormalities in Treatment and FU Periods
Description: Vital signs include supine and standing systolic blood pressure (SBP) [millimeters of mercury (mmHg)]: <90, >180, increase and decrease from baseline of >=30; Supine and standing diastolic blood pressure (DBP) (mmHg): Increase and decrease from baseline >=20; Standing heart rate (>120 beats per minute); Orthostatic SBP (>=20); Orthostatic DBP (>=10); Orthostatic hypotension (SBP >=20 and DBP >=10, SBP >=20 or DBP >=10).
Time Frame: Treatment period: Up to Day 14; FU period: Day 15 to 42
Population: Safety Set included all participants who were administered IP in treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period: SAGE-217 Matched Placebo | Treatment Period: SAGE-217 20 mg | Treatment Period: SAGE-217 30 mg | FU Period: SAGE-217 Matched Placebo | FU Period: SAGE-217 20 mg | FU Period: SAGE-217 30 mg
Number analyzed (Participants) | 190 | 188 | 192 | 190 | 188 | 192
Participants | 0 | 0 | 0 | 0 | 0 | 0

25. Secondary Outcome: Number of Participants With Clinically Significant Vital Sign Abnormalities in Extended FU Period
Description: Vital signs include supine and standing SBP [mmHg]: <90, >180, increase and decrease from baseline of >=30; Supine and standing DBP (mmHg): Increase and decrease from baseline >=20; Standing heart rate (>120 beats per minute); Orthostatic SBP (>=20); Orthostatic DBP (>=10); Orthostatic hypotension (SBP >=20 and DBP >=10, SBP >=20 or DBP >=10).
Time Frame: Extended FU Period: Day 43 to 182
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Extended FU Period: SAGE-217 Matched Placebo | Extended FU Period: SAGE-217 20 mg | Extended FU Period: SAGE-217 30 mg
Number analyzed (Participants) | 129 | 127 | 131
Participants | 0 | 0 | 0

26. Secondary Outcome: Number of Participants With Clinically Significant Electrocardiogram (ECG) Abnormalities in Treatment and FU Periods
Description: Supine 12-lead ECGs were performed in triplicate and the standard intervals (heart rate, PR, QRS, QT, and corrected QT interval by Fridericia [QTcF]) as well as any rhythm abnormalities were recorded. Criteria for clinically significant ECG abnormalities included QTcF interval (msec)- females: >450 to 480, male: >450 to 470, females: >480 to 500, male: >470 to 500 or >500.
Time Frame: Treatment period: Up to Day 14; FU period: Day 15 to 42
Population: Safety Set included all participants who were administered IP in treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period: SAGE-217 Matched Placebo | Treatment Period: SAGE-217 20 mg | Treatment Period: SAGE-217 30 mg | FU Period: SAGE-217 Matched Placebo | FU Period: SAGE-217 20 mg | FU Period: SAGE-217 30 mg
Number analyzed (Participants) | 190 | 188 | 192 | 190 | 188 | 192
Participants | 0 | 0 | 0 | 0 | 0 | 0

27. Secondary Outcome: Number of Participants With Clinically Significant ECG Abnormalities in Extended FU Period
Description: Supine 12-lead ECGs were performed in triplicate and the standard intervals (heart rate, PR, QRS, QT, and QTcF) as well as any rhythm abnormalities were recorded. Criteria for clinically significant ECG abnormalities included QTcF interval (msec)- females: >450 to 480, male: >450 to 470, females: >480 to 500, male: >470 to 500 or >500.
Time Frame: Extended FU Period: Day 43 to 182
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Extended FU Period: SAGE-217 Matched Placebo | Extended FU Period: SAGE-217 20 mg | Extended FU Period: SAGE-217 30 mg
Number analyzed (Participants) | 129 | 127 | 131
Participants | 0 | 0 | 0

28. Secondary Outcome: Number of Participants With Suicidal Ideation or Behavior Assessed Using the Columbia Suicide Severity Rating Scale (C-SSRS) in Double-blind Treatment Period at Day 42
Description: Suicidality was monitored during the study using the C-SSRS scale. The C-SSRS includes 'yes' or 'no' responses for 5 questions for assessment of suicidal ideation and behavior. Any suicidal behavior: When response is "yes" for any these questions- actual attempt to suicide, engaged in non-suicidal self-injurious behavior, interrupted attempt, aborted attempt, preparatory acts. Any suicidal ideation: When response is "yes" for any of these questions- wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent to suicide.
Time Frame: Day 42
Population: Safety Set included all participants who were administered IP in treatment period. This outcome measure was planned to be assessed for all participants in the Safety Set by summarizing and reporting data for treatment and FU periods combined together as double-blind treatment period.
Measure: Count of Participants; unit: Participants
Groups:
- Double-blind Treatment Period: SAGE-217 Matched Placebo: Participants self-administered SAGE-217 matched placebo capsules, orally, once daily in the evening with food for 14 days and were followed up for 28 days.
- Double-blind Treatment Period: SAGE-217 20 mg: Participants self-administered SAGE-217 20 mg capsules, orally, once daily in the evening with food for 14 days and were followed up for 28 days.
- Double-blind Treatment Period: SAGE-217 30 mg: Participants self-administered SAGE-217 30 mg capsules, orally, once daily in the evening with food for 14 days and were followed up for 28 days.
Arm/Group | Double-blind Treatment Period: SAGE-217 Matched Placebo | Double-blind Treatment Period: SAGE-217 20 mg | Double-blind Treatment Period: SAGE-217 30 mg
Number analyzed (Participants) | 190 | 188 | 192
Participants | 12 | 11 | 11

29. Secondary Outcome: Number of Participants With Suicidal Ideation or Behavior Assessed Using the Columbia Suicide Severity Rating Scale (C-SSRS) in Extended FU Period at Day 182
Description: as for outcome 28
Time Frame: Day 182
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Extended FU Period: SAGE-217 Matched Placebo | Extended FU Period: SAGE-217 20 mg | Extended FU Period: SAGE-217 30 mg
Number analyzed (Participants) | 129 | 127 | 131
Participants | 9 | 6 | 3

30. Secondary Outcome: Change From Baseline in the 20-item Physician Withdrawal Checklist (PWC-20) Total Score
Description: The PWC-20 was used to monitor for the presence of potential withdrawal symptoms following discontinuation of SAGE-217. The PWC-20 was made up of a list of 20 symptoms (loss of appetite, nausea-vomiting, diarrhea, anxiety-nervousness, irritability, dysphoric mood-depression, insomnia, fatigue-lethargy-lack of energy, poor coordination, restlessness-agitation, diaphoresis, tremor-tremulousness, dizziness-lightheadedness, headaches, muscle aches or stiffness, weakness, increased acuity [sound, smell, touch, pain], paresthesia, difficulty concentrating and remembering, depersonalization-derealization) that were rated on a scale of 0 (not present) to 3 (severe). The PWC-20 total score was derived as the sum of individual item scores, which ranges from 0 (not present) to 60 (severe). Higher scores indicate more severe withdrawal. A negative change from baseline indicates less severe withdrawal.
Time Frame: Baseline, Days 15, 18, and 21
Population: Safety Set included all participants who were administered IP. Here, "Overall number of participants analyzed" is the number of participants with data available for analyses. "Number analyzed" is the number of participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SAGE-217 Matched Placebo | SAGE-217 20 mg | SAGE-217 30 mg
Number analyzed (Participants) | 169 | 175 | 172
score on a scale
  Change from Baseline at Day 15: number analyzed (Participants) | 167 | 175 | 172
  Change from Baseline at Day 15 | -5.407 (7.0047) | -5.370 (7.5424) | -5.699 (7.7363)
  Change from Baseline at Day 18: number analyzed (Participants) | 163 | 174 | 168
  Change from Baseline at Day 18 | -6.128 (6.9928) | -5.421 (7.0046) | -5.917 (7.7158)
  Change from Baseline at Day 21: number analyzed (Participants) | 169 | 171 | 168
  Change from Baseline at Day 21 | -5.623 (7.2786) | -6.136 (7.2765) | -5.961 (7.0005)

ADVERSE EVENTS:
Time Frame: Treatment period: Up to 14 days; FU period: Day 15 to 42; Extended FU Period: Day 43 to 182
Description: Treatment and FU periods: Safety Set included all participants who were administered IP. FU period: Safety Set included all participants who were administered IP in treatment period. Extended FU period: Extended FU Safety Set included all participants in the Safety Set of treatment period who consented or reconsented to participate in the study in the 6-month FU period. The AE data were collected and reported period-wise.
Arm/Group | Treatment Period: SAGE-217 Matched Placebo | Treatment Period: SAGE-217 20 mg | Treatment Period: SAGE-217 30 mg | FU Period: SAGE-217 Matched Placebo | FU Period: SAGE-217 20 mg | FU Period: SAGE-217 30 mg | Extended FU Period: SAGE-217 Matched Placebo | Extended FU Period: SAGE-217 20 mg | Extended FU Period: SAGE-217 30 mg
All-Cause Mortality (participants affected / at risk) | 0/190 | 0/188 | 0/192 | 0/190 | 0/188 | 0/192 | 0/129 | 1/127 | 0/131
Serious Adverse Events (participants affected / at risk) | 0/190 | 0/188 | 2/192 | 1/190 | 1/188 | 1/192 | 1/129 | 3/127 | 1/131
Other Adverse Events (participants affected / at risk) | 43/190 | 53/188 | 60/192 | 0/190 | 0/188 | 0/192 | 0/129 | 0/127 | 0/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Period: SAGE-217 Matched Placebo (N=190) | Treatment Period: SAGE-217 20 mg (N=188) | Treatment Period: SAGE-217 30 mg (N=192) | FU Period: SAGE-217 Matched Placebo (N=190) | FU Period: SAGE-217 20 mg (N=188) | FU Period: SAGE-217 30 mg (N=192) | Extended FU Period: SAGE-217 Matched Placebo (N=129) | Extended FU Period: SAGE-217 20 mg (N=127) | Extended FU Period: SAGE-217 30 mg (N=131)
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Drug abuse (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mania (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Toxic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Period: SAGE-217 Matched Placebo (N=190) | Treatment Period: SAGE-217 20 mg (N=188) | Treatment Period: SAGE-217 30 mg (N=192) | FU Period: SAGE-217 Matched Placebo (N=190) | FU Period: SAGE-217 20 mg (N=188) | FU Period: SAGE-217 30 mg (N=192) | Extended FU Period: SAGE-217 Matched Placebo (N=129) | Extended FU Period: SAGE-217 20 mg (N=127) | Extended FU Period: SAGE-217 30 mg (N=131)
Headache (Nervous system disorders) | 14 | 21 | 12 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 7 | 14 | 11 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 8 | 11 | 13 | 0 | 0 | 0 | 0 | 0 | 0
Sedation (Nervous system disorders) | 6 | 11 | 9 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 10 | 11 | 12 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 9 | 10 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (Gastrointestinal disorders) | 5 | 3 | 13 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for non-commercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/75/NCT03672175/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-12): https://cdn.clinicaltrials.gov/large-docs/75/NCT03672175/SAP_001.pdf